CLINICAL TRIAL: NCT06963450
Title: Clinical Investigation of the Smartphone App neoSCB to Perform Neonatal Jaundice Screening in Newborn Babies
Brief Title: NeoSCB App for Screening Jaundice in Newborns
Acronym: neoSCB
Status: Recruiting | Type: Observational
Sponsor: University College, London (Other)
Collaborators: University College London Hospitals (Other)
Responsible Party: Sponsor
Other Study IDs: 157238; NIHR205460 (Other Grant/Funding Number: National Institute for Health and Care Research)
Record Dates: First submitted 2025-05-06; First posted 2025-05-09 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Neonatal Jaundice
Keywords: screening; newborn babies; mobile app; neonatal jaundice
MeSH Terms: conditions — Jaundice, Neonatal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Newborns: Term newborn babies with postnatal age 9 to 28 days
  Interventions: Diagnostic Test: Taking photos of a baby's eye

INTERVENTIONS:
Diagnostic Test: Taking photos of a baby's eye — Taking photos of a baby's eye and using the color of the sclera to estimate the bilirubin level, which determines if the baby is significantly jaundiced.

SUMMARY:
About 60% of babies born after 36 weeks of pregnancy have jaundice during the first two weeks of life. Due to the accumulation of bilirubin in the bloodstream, jaundiced babies appear yellow, which allows healthcare professionals to visually identify significantly jaundiced babies. They will be referred for a blood test to determine if the bilirubin level is so high that treatment such as phototherapy, or more intensive help is required. Left untreated or treatment delayed, jaundice can potentially result in serious brain damage and even death (rare). However, visual inspection of jaundiced babies is inaccurate, often need to unnecessary referrals to hospital blood tests. We have developed the "neoSCB" smartphone app, which accurately detects significant jaundice by taking photographs of the baby's sclera (white part of an eye) and analysing its yellowness using a diagnostic algorithm. The neoSCB app has previously been validated in Ghana involving over 700 newborn babies. In this new study, we will recruit 405 newborn babies with a range of jaundice levels to validate an optimised diagnostic algorithm following our latest research. Two existing commercial screening devices will also be used to investigate whether the app delivers a similar accuracy, at a fraction of the cost. We will enhance the usability of the app and add new features following feedback from patients and healthcare professionals. A health economic study will be conducted to evaluate the economic benefits to the NHS.

ELIGIBILITY:
Inclusion Criteria:

* Term newborn babies with and without jaundice (postnatal age 0 day to 28 days)

Exclusion Criteria:

* Newborn babies who are clinically unwell and require urgent medical attention, and babies who have received phototherapy recently

Max Age: 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Newborn babies are all recruited from UCL Hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 405 (Estimated)
Dates: Start 2025-09-23 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Total serum bilirubin | The measurement of total serum bilirubin should take less than 10 minutes.
  Total serum bilirubin is measured by taking a blood sample from the newborn baby. It is a standard way to assess how jaundiced the baby is and if a treatment is necessary.
Scleral-conjunctival bilirubin | The measurement of scleral-conjunctival bilirubin should take less than 5 minutes.
  Scleral-conjunctival bilirubin is estimated from digital photos of the baby's eye, based on the color of the sclera. It is a non-invasive way to estimate bilirubin, allowing the assessment of how jaundiced a baby is and whether a confirmatory blood test is required.

CONTACTS AND LOCATIONS:
Overall Officials: Judith Meek, MBBS, Principal Investigator — UCL Hospitals
Locations (1):
- UCL Hospitals, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
The data include partial face photos of newborn babies which are personal information and cannot be shared due to privacy concern.

REFERENCES:
- [Background] Leung TS, Outlaw F, MacDonald LW, Meek J. Jaundice Eye Color Index (JECI): quantifying the yellowness of the sclera in jaundiced neonates with digital photography. Biomed Opt Express. 2019 Feb 14;10(3):1250-1256. doi: 10.1364/BOE.10.001250. eCollection 2019 Mar 1. PMID 30891343
- [Background] Leung TS, Kapur K, Guilliam A, Okell J, Lim B, MacDonald LW, Meek J. Screening neonatal jaundice based on the sclera color of the eye using digital photography. Biomed Opt Express. 2015 Oct 23;6(11):4529-38. doi: 10.1364/BOE.6.004529. eCollection 2015 Nov 1. PMID 26601015
- [Background] Enweronu-Laryea C, Leung T, Outlaw F, Brako NO, Insaidoo G, Hagan-Seneadza NA, Ani-Amponsah M, Nixon-Hill M, Meek J. Validating a Sclera-Based Smartphone Application for Screening Jaundiced Newborns in Ghana. Pediatrics. 2022 Jul 1;150(1):e2021053600. doi: 10.1542/peds.2021-053600. PMID 35656782
- [Background] Outlaw F, Nixon M, Odeyemi O, MacDonald LW, Meek J, Leung TS. Smartphone screening for neonatal jaundice via ambient-subtracted sclera chromaticity. PLoS One. 2020 Mar 2;15(3):e0216970. doi: 10.1371/journal.pone.0216970. eCollection 2020. PMID 32119664
- See also: Website providing background information and methodology of the neoSCB screening app — http://www.detect-jaundice.org